CLINICAL TRIAL: NCT00999921
Title: A Single Blinded Randomized Controlled Trial of the Comparative Effects of Tamoxifen and Evening Primrose Oil in Premenopausal Non-high Risk Patients With Benign Breast Disease With Respect to the Estrogen Receptor Status.
Brief Title: Effects of Tamoxifen in Premenopausal Women With Benign Breast Disease Not at High-Risk of Developing Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College and Hospital Kolkata (Other)
Responsible Party: Principal Investigator, Md Tanveer Adil, Resident, Medical College and Hospital Kolkata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSVP-107/08
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-04

CONDITIONS: Benign Breast Disease; Fibrocystic Disease of Breast; Fibroadenoma; Mastalgia
Keywords: Fibrocystic Breast Disease; Fibroadenoma; Mastalgia
MeSH Terms: conditions — Cystic Fibrosis; Fibrocystic Breast Disease; Fibroadenoma; Mastodynia | interventions — Tamoxifen; evening primrose oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamoxifen (Experimental): 10 mg once daily from 5th day to 25th day of menstrual cycle for 3 months
  Interventions: Drug: Tamoxifen
- Evening Primrose Oil (Experimental): 1000 mg daily for 3 months
  Interventions: Drug: Evening Primrose Oil

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen is given at 10 mg once daily between Day 5 and Day 25 of menstrual cycle for 3 cycles.
  Arms: Tamoxifen
Drug: Evening Primrose Oil — Evening Primrose Oil is given at 1000 mg two times daily for 3 months.
  Arms: Evening Primrose Oil

SUMMARY:
The purpose of the study is to determine the efficacy and relapse rate of low dose, short duration treatment with tamoxifen in benign breast disease amenable to hormonal therapy with respect to etiology and estrogen receptor status and to realize its side-effects and cost of therapy.

To do a comparative analysis of the results with evening primrose oil which is one of the first line management in benign breast disease.

DETAILED DESCRIPTION:
Benign breast disease is frequently encountered in female patients, a significant proportion of who are premenopausal women. Established methods of treatment do not yield significant results. This is not only a social burden but also entails high economic cost. As such the quality of life of these patients is a matter of concern for both the patients and their families and to attending physicians. Reported effects of tamoxifen on benign breast disease in premenopausal non high risk patients are scarce. Moreover published data has not yet revealed association of estrogen receptors in different benign breast lesions.The variability of response and its relation with estrogen receptor status is still a field of active investigation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical, Radiographic and Histological diagnosis of Benign Breast Disease.
* Benign Breast disease amenable to hormonal therapy.

Exclusion Criteria:

* Postmenopausal women.
* Premenopausal women with pregnancy or other contraindications to tamoxifen.
* Girls less than 16 years.
* Very large lesions which require surgery for cosmesis.
* High risk breast lesions like epitheliosis, atypia or atypical hyperplasia on histopathology or susceptible lesions prone to develop malignancy.
* Lesions like duct ectasia where hormone therapy is not likely to be of benefit.
* Inflammatory lesions which are amenable to antibiotic therapy or surgical drainage for treatment.
* Patients unwilling to undergo treatment.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2008-01; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Md Tanveer Adil, Principal Investigator — Resident, Department of Surgery, Medical College and Hospital, Kolkata; Rumana Rahman, Study Director — Resident, Department of Gynaecology and Obstetrics, Medical College and Hospital, Kolkata; Soumen Das, Study Director — Resident, Department of Surgery, Medical College and Hospital, Kolkata; Sudip Sarkar, Study Director — Resident, Department of Surgery, Medical College and Hospital, Kolkata; Rupesh Kumar, Study Director — Resident, Department of Surgery, Medical College and Hospital, Kolkata; Utpal De, Study Chair — Professor, Department of Surgery, Medical College and Hospital, Kolkata
Locations (1):
- Department of Surgery, Medical College, Kolkata, Kolkata, West Bengal, India

REFERENCES:
- [Background] Srivastava A, Mansel RE, Arvind N, Prasad K, Dhar A, Chabra A. Evidence-based management of Mastalgia: a meta-analysis of randomised trials. Breast. 2007 Oct;16(5):503-12. doi: 10.1016/j.breast.2007.03.003. Epub 2007 May 16. PMID 17509880
- [Background] Allegra JC, Lippman ME, Green L, Barlock A, Simon R, Thompson EB, Huff KK, Griffin W. Estrogen receptor values in patients with benign breast disease. Cancer. 1979 Jul;44(1):228-31. doi: 10.1002/1097-0142(197907)44:13.0.co;2-0. PMID 455247
- [Background] Hurst JL, Mega JF, Hogg JP. Tamoxifen-induced regression of breast cysts. Clin Imaging. 1998 Mar-Apr;22(2):95-8. doi: 10.1016/s0899-7071(97)00076-4. PMID 9543585
- [Background] Tan-Chiu E, Wang J, Costantino JP, Paik S, Butch C, Wickerham DL, Fisher B, Wolmark N. Effects of tamoxifen on benign breast disease in women at high risk for breast cancer. J Natl Cancer Inst. 2003 Feb 19;95(4):302-7. doi: 10.1093/jnci/95.4.302. PMID 12591986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Premenopausal women with Benign Breast Disease and who belong to non-high risk group for breast cancer were included in the study
Pre-assignment Details: Postmenopausal women, premenopausal women with pregnancy or other contraindications to tamoxifen, girls less than 15 years, very large lesions, high risk patients with epitheliosis, atypia or atypical hyperplasia or prone to develop malignancy and patients unwilling to undergo treatment were excluded from the study
Groups:
- Tamoxifen: Tamoxifen 10 mg OD from 5th day to 25th day of menstrual cycle for 3 months
- Evening Primrose Oil: Evening Primrose Oil 1000 mg daily for 3 months
Period: Overall Study
Arm/Group | Tamoxifen | Evening Primrose Oil
Started | 127 | 129
Completed | 117 | 110
Not Completed | 10 | 19
Not completed — Lost to Follow-up | 10 | 19

BASELINE CHARACTERISTICS:
Groups:
- Tamoxifen: Tamoxifen was administered at a dose of 10 mg once daily ffrom 5th day to 25 th day of menstrual cycle for 3 months
- Evening Primrose Oil: Evening Primrose Oil was administered at a dose of 1000 mg daily for 3 months
- Total: Total of all reporting groups
Arm/Group | Tamoxifen | Evening Primrose Oil | Total
Number analyzed (Participants) | 127 | 129 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 124 | 127 | 251
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.38 (4.2) | 25.16 (3.8) | 25.27 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 129 | 256
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 127 | 129 | 256

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Analysed for Reduction in Lump Size ( 60% Reduction in Lump Size Considered to be a Satisfactory Response)
Description: Ultrasonography of the breast was used to ascertain the lump size at the beginning of therapy and a repeat Ultrasonography of breast was done after 3 months at the end of the proposed therapy to record the posttreatment lump size by the same operator. The difference between the two findings were recorded and noted and a 60% or more reduction in the size of the lump was considered as a satisfactory response.
Time Frame: 3 months
Population: 102(out of 127) patients receiving Tamoxifen and 99(out of 129) receiving Evening Primrose Oil were assessed for reduction in lump size. The remaining patients had mastalgia with no lump, hence were excluded from this assessment. A 60% or more reduction in lump size after completion of the therapy was considered as a satisfactory response.
Measure: Number; unit: participants
Groups:
- Tamoxifen: Tamoxifen at a dose of 10 mg once daily from 5th day to 25th day of menstrual cycle for 3 months
- Evening Primrose Oil: Evening Primrose Oil at a dose of 1000 mg once daily for 3 months
Arm/Group | Tamoxifen | Evening Primrose Oil
Number analyzed (Participants) | 102 | 99
participants
  Fibroadenosis (total number) | 63 | 61
  Fibroadenosis (60% or more reduction in size) | 54 | 14
  Fibroadenosis (less than 60% reduction in size) | 9 | 47
  Fibroadenoma (total number) | 39 | 38
  Fibroadenoma (60% or more reduction in size) | 4 | 0
  Fibroadenoma (less than 60% reduction in size) | 35 | 38

2. Primary Outcome: Number of Participants Analysed for Reduction in Mastalgia (Cardiff Breast Pain Score).
Description: All patients were categorized as Grade 0 for no pain, grade 1 for mild pain, grade 2 for moderate pain, Grade 3 for severe pain. Therapeutic response to mastalgia was expressed in terms of Cardiff Breast Pain Score (CBS) where CBS I = excellent response with no pain, CBS II = substantial response, CBS III = poor response and CBS IV = no response
Time Frame: 3 months
Population: 88 patients treated with Tamoxifen and 47 patients treated with Evening Primrose Oil were assessed for Cardiff Breast Pain Score. Patients with fibroadenomas and those with Grade 0 pain at the beginning of therapy were excluded from this analysis.
Measure: Number; unit: participants
Groups:
- Tamoxifen: Tamoxifen administered at a dose of 10 mg once daily from 5th day to 25th day of menstrual cycle for 3 months
- Evening Primrose Oil: Evening Primrose Oil was administered at a dose of 1000 mg once daily for 3 months
Arm/Group | Tamoxifen | Evening Primrose Oil
Number analyzed (Participants) | 88 | 47
participants
  CBS I (excellent response) | 71 | 10
  CBS II (substantial response) | 13 | 15
  CBS III (poor response) | 3 | 11
  CBS IV (no response) | 1 | 11

3. Secondary Outcome: Number of Participants Analysed for Response of Cyclical Mastalgia (Good Response Was Defined as Disappearance of Mastalgia)
Description: All patients who had an increase in breast pain in the "perimenstrual period" were designated as having cyclical mastalgia. Response was assessed following treatment in terms of either persistence of cyclical mastalgia after 3 months of treatment or disappearance of cyclical mastalgia
Time Frame: 3 months
Population: 114 patients were identified as having cyclical mastalgia of whom 58 patients(37 fibroadenosis, 3 fibroadenonomas and 18 mastalgias with no lump) received Tamoxifen and 56 (36 fibroadenosis, 3 fibroadenomas and 17 mastalgias with no lump) received Evening Primrose Oil for 3 months. Good response was defined as disappearance of cyclical mastalgia.
Measure: Number; unit: participants
Groups:
- Tamoxifen: Tamoxifen was administered at a dose of 10 mg once daily from 5th day to 25th day of menstrual cycle for 3 months
Arm/Group | Tamoxifen | Evening Primrose Oil
Number analyzed (Participants) | 58 | 56
participants
  Fibroadenosis(total number) | 37 | 36
  Fibroadenosis (good response) | 30 | 11
  Fibroadenosis (poor response) | 7 | 25
  Fibroadenoma (total number) | 3 | 3
  Fibroadenoma (good response) | 3 | 1
  Fibroadenoma (poor response) | 0 | 2
  Mastalgia with no lump (total number) | 18 | 17
  Mastalgia with no lump (good response) | 17 | 3
  Mastalgia with no lump (poor response) | 1 | 14

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed at 3 months after completion of therapy, after a 3 month followup and at 6 month followup
Description: Major adverse effect = Menstrual Irregularity,
  Minor adverse effects = 1) Hot flushes 2) Nausea and vomiting 3) Mood changes
  Presence of major or minor adverse effect at any period of followup was considered as an adverse effect of the total number of participants in the respective arm of the study.
Arm/Group | Tamoxifen | Evening Primrose Oil
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/129
Other Adverse Events (participants affected / at risk) | 82/127 | 0/129
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen (N=127) | Evening Primrose Oil (N=129)
Hot Flushes (Skin and subcutaneous tissue disorders) | 59 (59) | 0 (0) — Hot flushes was objectively assessed as a feeling of intense heat with or without sweating and rapid heart beat
Nausea (Gastrointestinal disorders) | 19 (19) | 0 (0) — Nausea was noted as a feeling of discomfort in upper abdomen with an involuntary urge to vomit
Mood Changes (Psychiatric disorders) | 4 (4) | 0 (0) — Mood changes were defined as rapid or extreme change in mood

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes